CLINICAL TRIAL: NCT01842269
Title: Open Label, Randomized, Multi-center, Phase 4 Trial to Evaluate the Efficacy and Safety of My-Rept® Tablet(Mycophenolate Mofetil 500mg/Tab.) Versus My-Rept® Capsule(Mycophenolate Mofetil 250mg/Cap.) in Combination With Tacrolimus for 26 Weeks in Kidney Transplant Patients
Brief Title: Evaluate the Efficacy and Safety of My-Rept® Tablet vs. My-Rept® Capsule in Combination With Tacrolimus in Kidney Transplant Patients
Acronym: My-Rept_KT_P4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 223KTP12003
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Transplantation
Keywords: Mycophenolate Mofetil; MMF
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- My-Rept® Tablet (Experimental): My-Rept® Tablet, Mycophenolate Mofetil 500mg, orally
  Interventions: Drug: Mycophenolate Mofetil 500mg
- My-Rept® Capsule (Active Comparator): My-Rept® Capsule, Mycophenolate Mofetil 250mg, orally
  Interventions: Drug: Mycophenolate Mofetil 250mg

INTERVENTIONS:
Drug: Mycophenolate Mofetil 500mg
  Other Names: My-Rept® Tablet
  Arms: My-Rept® Tablet
Drug: Mycophenolate Mofetil 250mg
  Other Names: My-Rept® Capsule
  Arms: My-Rept® Capsule

SUMMARY:
Efficacy and Safety of My-Rept® Tablet(Mycophenolate Mofetil 500mg/Tab.) versus My-Rept® Capsule(Mycophenolate Mofetil 250mg/Cap.) in Combination with Tacrolimus in Kidney Transplant Patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 years or older.
2. Patient who receive primary or secondary kidney transplantation from living or brain-dead donor .
3. Patient who receive age 20 years or older donor.
4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Cold Ischemia Time > 30 hours.
2. Patient who receive HLA-identical donor.
3. Patient with dual kidney transplantation recipient or have history of other organ transplantation in past or current.
4. Patient who receive extra-renal solid organ or bone marrow stem cell transplantation.
5. Patient who receive kidney transplantation from non-heart beating cadaveric donor(organ donor after cardiac death
6. Patient who receive kidney transplantation from ABO blood type mismatching donor or lymphocyte cross matching (LCM) positive donor.
7. Patient with cancer within 5 years, except cured skin cancer patient(Squamous cell or basal cell carcinoma)
8. Positive in serology test(HIV, HBsAg, HCV) in recipients and/or donor.
9. Patient with Severe gastrointestinal disease in screening period by investigator's decision.
10. Patient with systemic severe infection requiring treatment (able to transplantation after completely disappear or is controlled infection)
11. Liver cirrhosis, clinically significant portal hypertension or other moderate to severe liver disease.
12. Defined by the following laboratory parameters before screening period

    1. One of liver function test(AST, ALT, ALP, Total Bilirubin)results increased more than 3 times upper limit of normal range
    2. WBC <2,500/mm3, Platelet <75,000/mm3
13. Acute (within 4 weeks) or chronic(need to treatments) allergic/hypersensitivity reaction in the history of Investigational drugs (ex, mycophenolate acid or tacrolimus, etc.) or additives.
14. Administration of other Investigational drugs and/or immunosuppressants within 28days before screening period (except allowed immunosuppressants in protocol)
15. Women in pregnant or breast-feeding or don't using adequate contraception.
16. Patient has conversation impairment because alcohol or drugs addiction history within 6months or mental illness, etc.
17. In investigator's judgment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Rate of efficacy failure | up to 26 weeks
  efficacy failure=acute rejection by kidney biopsy,graft loss, death

SECONDARY OUTCOMES:
Rate of acute rejection by kidney biopsy | up to 26 weeks
Survival with no graft loss | up to 26 weeks
eGFR(using by MDRD method) | up to 26 weeks
Number of Participants with Adverse Events | up to 26 weeks
  * Rate of adverse events
  * Evaluated safety parameters included: Physical examination, laboratory test, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Seun Kim, Ph. D, Principal Investigator — Severance Hospital
Locations (11):
- South Korea (11):
  - Maryknoll Medical Center, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Wonkwang University School of Medical & Hospital, Iksan
  - Chunbuk National University Hospital, Jeonju
  - Bundang CHA Medical Center, Seongnam
  - Gangnam Severance Hospital, Seoul
  - Kandong Sacred Heart Hospital, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwan
  - Ulsan University Hospital, Ulsan